CLINICAL TRIAL: NCT01854658
Title: A Randomized, Double-Blind (Test Products and Placebo), Chronic Dosing (24 Weeks), Placebo-Controlled, Parallel Group, Multi-Center Study to Assess the Efficacy and Safety of PT003, PT005, and PT001 in Subjects With Moderate to Very Severe COPD, Compared With Placebo
Brief Title: Multi-Center Study to Assess the Efficacy and Safety of PT003, PT005, and PT001 in Subjects With Moderate to Very Severe COPD (PINNACLE 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT003007-00
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FF MDI (PT005) (Experimental): FF MDI administered as two puffs BID
  Interventions: Drug: FF MDI (PT005)
- GP MDI (PT001) (Experimental): GP MDI administered as two puffs BID
  Interventions: Drug: GP MDI (PT001)
- GFF MDI (PT003) (Experimental): GFF MDI administered as two puffs BID
  Interventions: Drug: GFF MDI (PT003)
- Placebo MDI (Placebo Comparator): Inhaled placebo administered as two puffs BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFF MDI (PT003) — GFF MDI administered as two puffs BID
  Other Names: glycopyrrolate/formoterol fumarate metered-dose inhaler; (GFF MDI)
  Arms: GFF MDI (PT003)
Drug: GP MDI (PT001) — GP MDI administered as two puffs BID
  Other Names: glycopyrrolate metered dose inhaler (GP MDI)
  Arms: GP MDI (PT001)
Drug: FF MDI (PT005) — FF MDI administered as two puffs BID
  Other Names: formoterol fumarate metered dose inhaler (FF MDI)
  Arms: FF MDI (PT005)
Drug: Placebo
  Arms: Placebo MDI

SUMMARY:
This is a multicenter, randomized, double-blind, parallel group, chronic-dosing (24 weeks), placebo-controlled study to assess the efficacy and safety of Glycopyrrolate (GP and Formoterol Fumarate (FF) combination metered-dose inhaler (MDI) (GFF; PT003), GP MDI (PT001), and FF MDI (PT005) compared with Placebo MDI in subjects with moderate to very severe COPD.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects at least 40 years of age and no older than 80 at Visit 1.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Subjects with FEV1/FVC ratio of <0.70 and FEV1 <80% predicted normal and ≥750 mL if FEV1 <30% of predicted normal value.
* Subjects willing and, in the opinion of the investigator, able to adjust current COPD therapy as required by the protocol

Key Exclusion Criteria:

* Significant diseases other than COPD, i.e. disease or condition which, in the opinion of the investigator, may put the patient at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study
* Current diagnosis of asthma or alpha-1 antitrypsin deficiency
* Other active pulmonary disease such as active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, idiopathic interstitial pulmonary fibrosis, primary pulmonary hypertension, or uncontrolled sleep apnea
* Hospitalized due to poorly controlled COPD within 3 months prior to screening or during the Screening Period
* Poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to screening or during the Screening Period
* Lower respiratory tract infections that required antibiotics within 6 weeks prior to screening or during the Screening Period
* Unstable ischemic heart disease, left ventricular failure, or documented myocardial infarction within 12 months of enrollment.
* Recent history of acute coronary syndrome, percutaneous coronary intervention, coronary artery bypass graft within the past three months
* Congestive heart failure (CHF NYHA Class III/IV)
* Clinically significant abnormal 12-lead ECG
* Abnormal liver function tests defined as AST, ALT, or total bilirubin ≥ 1.5 times upper limit of normal at Visit 1 and on repeat testing
* Cancer not in complete remission for at least five years
* History of hypersensitivity to β2-agonists, glycopyrronium or other muscarinic anticholinergics, lactose/milk protein or any component of the MDI

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1615 (Actual)
Dates: Start 2013-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Chair — Pearl Therapeutics, Inc.
Locations (113):
- United States (113):
  - Pearl Investigative Site, Birmingham, Alabama
  - Pearl Investigative Site, Florence, Alabama
  - Pearl Investigative Site, Jasper, Alabama
  - Pearl Investigative Site, Mobile, Alabama
  - Pearl Investigative Site, Fullerton, California
  - Pearl Investigative Site, Gold River, California
  - Pearl Investigative Site, Long Beach, California
  - Pearl Investigative Site, Los Angeles, California
  - Pearl Investigative Site, Mission Hills, California
  - Pearl Investigative Site, Newport Beach, California
  - Pearl Investigative Site, North Hollywood, California
  - Pearl Investigative Site, Northridge, California
  - Pearl Investigative Site, Rancho Mirage, California
  - Pearl Investigative Site, Rialto, California
  - Pearl Investigative Site, Rolling Hills Estates, California
  - Pearl Investigative Site, San Diego, California
  - Pearl Investigative Site, Santa Monica, California
  - Pearl Investigative Site, Stockton, California
  - Pearl Investigative Site, Torrance, California
  - Pearl Investigative Site, Wildomar, California
  - Pearl Investigative Site, Centennial, Colorado
  - Pearl Investigative Site, Boynton Beach, Florida
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Hialeah, Florida
  - Pearl Investigative Site, Jacksonville, Florida
  - Pearl Investigative Site, Kissimmee, Florida
  - Pearl Investigative Site, Melbourne, Florida
  - Pearl Investigative Site, Miami, Florida
  - Pearl Investigative Site, New Port Richey, Florida
  - Pearl Investigative Site, Orlando, Florida
  - Pearl Investigative Site, Ormond Beach, Florida
  - Pearl Investigative Site, Port Orange, Florida
  - Pearl Investigative Site, Sanford, Florida
  - Pearl Investigative Site, Sebring, Florida
  - Pearl Investigative Site, Tamarac, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Lawrenceville, Georgia
  - Pearl Investigative Site, Norcross, Georgia
  - Pearl Investigative Site, Smyrna, Georgia
  - Pearl Investigative Site, Elk Grove, Illinois
  - Pearl Investigative Site, Normal, Illinois
  - Pearl Investigative Site, Peoria, Illinois
  - Pearl Investigative Site, Evansville, Indiana
  - Pearl Investigative Site, Franklin, Indiana
  - Pearl Investigative Site, Lafayette, Indiana
  - Pearl Investigative Site, South Bend, Indiana
  - Pearl Investigative Site, Council Bluffs, Iowa
  - Pearl Investigative Site, Hazard, Kentucky
  - Pearl Investigative Site, Louisville, Kentucky
  - Pearl Investigative Site, Paducah, Kentucky
  - Pearl Investigative Site, Lake Charles, Louisiana
  - Pearl Investigative Siteq, Baltimore, Maryland
  - Pearl Investigative Site, Columbia, Maryland
  - Pearl Investigative Site, Haverhill, Massachusetts
  - Pearl Investigative Site, North Dartmouth, Massachusetts
  - Pearl Investigative Site, Ann Arbor, Michigan
  - Pearl Investigative Site, Fridley, Minnesota
  - Pearl Investigative Site, Minneapolis, Minnesota
  - Pearl Investigative Site, Rochester, Minnesota
  - Pearl Investigative Site, Saint Charles, Missouri
  - Pearl Investigative Site, St Louis, Missouri
  - Pearl Investigative Site, Fremont, Nebraska
  - Pearl Investigative Site, Omaha, Nebraska
  - Pearl Investigative Site, Henderson, Nevada
  - Pearl Investigative Site, Newington, New Hampshire
  - Pearl Investigative Site, Cedar Knolls, New Jersey
  - Pearl Investigative Site, Marlton, New Jersey
  - Pearl Investigative Site, Buffalo, New York
  - Pearl Investigative Site, New York, New York
  - Pearl Investigative Site, Rochester, New York
  - Pearl Investigative Site, Boone, North Carolina
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Hendersonville, North Carolina
  - Pearl Investigative Site, Raleigh, North Carolina
  - Pearl Investigative Site, Winston-Salem, North Carolina
  - Pearl Investigative Site, Akron, Ohio
  - Pearl Investigative Site, Canton, Ohio
  - Pearl Investigative Site, Cincinnati, Ohio
  - Pearl Investigative Site, Columbus, Ohio
  - Pearl Investigative Site, Willoughby, Ohio
  - Pearl Investigative Site, Oklahoma City, Oklahoma
  - Pearl Investigative Site, Tulsa, Oklahoma
  - Pearl Investigative Site, Portland, Oregon
  - Pearl Investigative Site, Hershey, Pennsylvania
  - Pearl Investigative Site, Phoenixville, Pennsylvania
  - Pearl Investigative Site, Pittsburgh, Pennsylvania
  - Pearl Investigative Site, Anderson, South Carolina
  - Pearl Investigative Site, Charleston, South Carolina
  - Pearl Investigative Site, Easley, South Carolina
  - Pearl Investigative Site, Fort Mill, South Carolina
  - Pearl Investigative Site, Gaffney, South Carolina
  - Pearl Investigative Site, Greenville, South Carolina
  - Pearl Investigative Site, Rock Hill, South Carolina
  - Pearl Investigative Site, Seneca, South Carolina
  - Pearl Investigative Site, Spartanburg, South Carolina
  - Pearl Investigative Site, Nashville, Tennessee
  - Pearl Investigative Site, Arlington, Texas
  - Pearl Investigative Site, Beaumont, Texas
  - Pearl Investigative Site, Boerne, Texas
  - Pearl Investigative Site, Corsicana, Texas
  - Pearl Investigative Site, Dallas, Texas
  - Pearl Investigative Site, Fort Worth, Texas
  - Pearl Investigative Site, Houston, Texas
  - Pearl Investigative Site, San Antonio, Texas
  - Pearl Investigative Site, Tomball, Texas
  - Pearl Investigative Site, Waco, Texas
  - Pearl Investigative Site, Midlothian, Virginia
  - Pearl Investigative Site, Newport News, Virginia
  - Pearl Investigative Site, Richmond, Virginia
  - Pearl Investigative Site, Ricmond, Virginia
  - Pearl Investigative Site, Spokane, Washington
  - Pearl Investigative Site, Tacoma, Washington
  - Pearl Investigative Site, Bridgeport, West Virginia

REFERENCES:
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359
- [Derived] Martinez FJ, Lipworth BJ, Rabe KF, Collier DJ, Ferguson GT, Sethi S, Feldman GJ, O'Brien G, Jenkins M, Reisner C. Benefits of glycopyrrolate/formoterol fumarate metered dose inhaler (GFF MDI) in improving lung function and reducing exacerbations in patients with moderate-to-very severe COPD: a pooled analysis of the PINNACLE studies. Respir Res. 2020 May 25;21(1):128. doi: 10.1186/s12931-020-01388-y. PMID 32450869
- [Derived] Martinez FJ, Rabe KF, Lipworth BJ, Arora S, Jenkins M, Martin UJ, Reisner C. Glycopyrrolate/Formoterol Fumarate Metered Dose Inhaler Improves Lung Function versus Monotherapies in GOLD Category A Patients with COPD: Pooled Data from the Phase III PINNACLE Studies. Int J Chron Obstruct Pulmon Dis. 2020 Jan 9;15:99-106. doi: 10.2147/COPD.S229794. eCollection 2020. PMID 32021148
- [Derived] Martinez FJ, Fabbri LM, Ferguson GT, Orevillo C, Darken P, Martin UJ, Reisner C. Baseline Symptom Score Impact on Benefits of Glycopyrrolate/Formoterol Metered Dose Inhaler in COPD. Chest. 2017 Dec;152(6):1169-1178. doi: 10.1016/j.chest.2017.07.007. Epub 2017 Jul 16. PMID 28720336
- See also: PT003007-02 Protocol Amendment-FINAL-Redacted.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4151&filename=PT003007-02%20Protocol%20Amendment-FINAL-11Sept14_29June16_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 140 sites throughout the United States from July 2013 - February 2015. Study participation was a maximum of 32 weeks.
Pre-assignment Details: A multicenter, randomized, double-blind, parallel group, chronic dosing, active- and placebo-controlled study; each participant was randomized to receive 1 of 4 possible treatments over the course of a 24-week treatment period (With a randomization of 7:6:6:3 GFF MDI, GP MDI, FF MDI and Placebo MDI)
Groups:
- FF MDI (PT005): FF MDI 9.6 mcg administered as two puffs BID
- GP MDI (PT001): GP MDI 14.4 mcg administered as two puffs BID
- GFF MDI (PT003): GFF MDI 14.4/9.6 mcg administered as two puffs BID
Period: Overall Study
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI
Started | 439 | 440 | 512 | 224
Completed | 346 | 365 | 432 | 165
Not Completed | 93 | 75 | 80 | 59
Not completed — Protocol Violation | 6 | 2 | 2 | 1
Not completed — Physician Decision | 7 | 5 | 2 | 4
Not completed — Lost to Follow-up | 8 | 9 | 8 | 4
Not completed — Withdrawal by Subject | 28 | 21 | 29 | 15
Not completed — Protocol-specified criteria | 15 | 15 | 10 | 7
Not completed — Lack of Efficacy | 3 | 8 | 4 | 7
Not completed — Adverse Event | 21 | 14 | 23 | 19
Not completed — Administrative reasons | 5 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: 5 subjects participated in more than one Phase 3 Pearl study (a protocol violation) and had overlapping treatment exposure - these subjects were removed from the ITT and safety populations;
  1 subject participated in more than one Phase 3 Pearl study but did not have overlapping treatment exposure - this subject was removed from the ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI | Total
Number analyzed (Participants) | 437 | 439 | 510 | 223 | 1609
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (7.8) | 62.8 (8.4) | 62.8 (8.2) | 64.2 (8.7) | 62.9 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 197 | 238 | 98 | 723
  Male | 247 | 242 | 272 | 125 | 886

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1
Description: Change from baseline in morning pre-dose trough forced expiratory volume in 1 second (FEV1) at Week 24.
Time Frame: At Week 24
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI
Number analyzed (Participants) | 350 | 367 | 433 | 170
Liters | 0.061 [0.039 to 0.082] | 0.063 [0.041 to 0.084] | 0.116 [0.097 to 0.136] | 0.013 [-0.018 to 0.044]

2. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 Over 24 Weeks
Description: Change from baseline in morning pre-dose trough forced expiratory volume in 1 second (FEV1) over 24 weeks. FEV1 was assessed at multiple time points post-baseline, and a model-based average of all visits starting from Week 2 through week 24 inclusive was calculated. The change values reported in the table represent the change between the baseline and the average FEV1 post-baseline.
Time Frame: Over 24 weeks
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI
Number analyzed (Participants) | 434 | 434 | 503 | 216
Liters | 0.080 [0.064 to 0.095] | 0.082 [0.067 to 0.097] | 0.137 [0.123 to 0.151] | 0.008 [-0.014 to 0.030]

3. Secondary Outcome: Peak FEV1
Description: Peak change from baseline in FEV1 within 2 hours post-dosing at Week 24
Time Frame: At week 24
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI
Number analyzed (Participants) | 346 | 365 | 431 | 165
Liters | 0.268 [0.244 to 0.292] | 0.223 [0.199 to 0.247] | 0.350 [0.328 to 0.371] | 0.083 [0.048 to 0.117]

4. Secondary Outcome: St. George Respiratory Questionnaire (SGRQ) Score
Description: Change from baseline in the SGRQ total score at Week 24. The SGRQ is a disease-specific questionnaire, self-completed by participants, used to evaluate the effect of GFF MDI, FF MDI and GP MDI on health-related quality of life as compared to placebo in subjects with COPD. The scores range from 0 (minimum, best possible health status) to 100 (maximum, worst possible health status). The SGRQ contains 76 items grouped into three domains (symptoms, activity and impacts). Change from Baseline at a particular visit was calculated as the SGRQ total score at that visit minus Baseline. Change from Baseline in total score of -4 units or lower is considered as clinically meaningful improvement in quality of life.
Time Frame: 24 weeks
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI
Number analyzed (Participants) | 352 | 362 | 430 | 170
Scores on a scale | -2.3 [-3.5 to -1.1] | -2.2 [-3.4 to -1.0] | -3.0 [-4.1 to -1.8] | -1.2 [-3.0 to 0.5]

5. Secondary Outcome: Rescue Ventolin HFA Use
Description: Change from baseline in average daily rescue Ventolin HFA use over 24 weeks
Time Frame: 24 weeks
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Puffs / Day
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI
Number analyzed (Participants) | 437 | 438 | 510 | 223
Puffs / Day | -0.7 [-0.9 to -0.5] | -0.4 [-0.6 to -0.3] | -1.0 [-1.2 to -0.8] | 0.0 [-0.2 to 0.3]

6. Secondary Outcome: Onset of Action as Assessed by FEV1
Description: Defined as the first time-point using the 5- and 15-minute post dose measurements where the difference in FEV1 from Placebo was statistically significant
Time Frame: Day 1
Population: Intent-to-Treat population with evaluable data (no imputation) for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI
Number analyzed (Participants) | 375 | 371 | 429 | 179
Liters
  5 min post dose | 0.175 [0.163 to 0.188] | 0.052 [0.040 to 0.065] | 0.192 [0.180 to 0.204] | 0.006 [-0.012 to 0.024]
  15 min post dose | 0.212 [0.199 to 0.225] | 0.109 [0.096 to 0.122] | 0.237 [0.225 to 0.249] | 0.022 [0.003 to 0.040]
Statistical Analysis 1: Comparison: FF MDI (PT005) vs Placebo MDI; At 5 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: FF MDI (PT005) vs Placebo MDI; At 15 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 3: Comparison: GP MDI (PT001) vs Placebo MDI; At 5 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 4: Comparison: GP MDI (PT001) vs Placebo MDI; At 15 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 5: Comparison: GFF MDI (PT003) vs Placebo MDI; At 5 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 6: Comparison: GFF MDI (PT003) vs Placebo MDI; At 15 min post dose; Test type: Superiority or Other; p < 0.0001, ANCOVA

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious Adverse Events (SAEs) will be collected from the time the subject signs the informed consent form up to 14 days following the last dose of study drug.
Description: Safety population included all participants who were administered investigational drug; participants were included in safety population according to the investigational drug received
Arm/Group | FF MDI (PT005) | GP MDI (PT001) | GFF MDI (PT003) | Placebo MDI
Serious Adverse Events (participants affected / at risk) | 37/438 | 37/439 | 36/510 | 15/223
Other Adverse Events (participants affected / at risk) | 21/438 | 12/439 | 22/510 | 10/223
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF MDI (PT005) (N=438) | GP MDI (PT001) (N=439) | GFF MDI (PT003) (N=510) | Placebo MDI (N=223)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 9 (9) | 8 (8) | 4 (4)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extradural abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (3) | 3 (3) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac pacemaker insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF MDI (PT005) (N=438) | GP MDI (PT001) (N=439) | GFF MDI (PT003) (N=510) | Placebo MDI (N=223)
Nasopharyngitis (Infections and infestations) | 21 (21) | 12 (12) | 22 (22) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.